CLINICAL TRIAL: NCT00785928
Title: Phase 2, Dose-Ranging Study of Multiple Subcutaneous Doses of LY2127399 in Patients With Active Rheumatoid Arthritis Despite Ongoing Methotrexate Therapy
Brief Title: A Study for Patients With Active Rheumatoid Arthritis Despite Ongoing Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12409; H9B-MC-BCDH (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Experimental)
  Interventions: Drug: Placebo
- 1 mg LY2127399 (Experimental)
  Interventions: Biological: LY2127399
- 3 mg LY2127399 (Experimental)
  Interventions: Biological: LY2127399
- 10 mg LY2127399 (Experimental)
  Interventions: Biological: LY2127399
- 30 mg LY2127399 (Experimental)
  Interventions: Biological: LY2127399
- 60 mg LY2127399 (Experimental)
  Interventions: Biological: LY2127399
- 120 mg LY2127399 (Experimental)
  Interventions: Biological: LY2127399

INTERVENTIONS:
Biological: LY2127399 — Administered SC every 4 weeks over a 24-week period (Weeks 0, 4, 8, 12, 16, and 20).
  Arms: 1 mg LY2127399; 10 mg LY2127399; 120 mg LY2127399; 3 mg LY2127399; 30 mg LY2127399; 60 mg LY2127399
Drug: Placebo — Administered subcutaneously (SC) every 4 weeks over a 24-week period (Weeks 0, 4, 8, 12, 16, and 20).
  Arms: Placebo

SUMMARY:
To assess the efficacy of LY2127399 versus placebo using American College of Rheumatology (ACR)50 response scale at 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Women must not be at risk to become pregnant during study participation
* Diagnosis of Rheumatoid Arthritis (RA)
* Current, regular use of Methotrexate, at a stable dose
* Other criteria to be reviewed by study doctor

Exclusion Criteria:

* Use of excluded medications(reviewed by study doctor)
* Have not failed biologic tumor necrosis factor-alpha (TNF-α) inhibitor therapy
* Have had recent or ongoing infection which, in the opinion of the study doctor put patient at an unacceptable risk for participation in the study
* Evidence of tuberculosis
* Have systemic inflammatory condition other than RA, such as juvenile RA, Crohn's disease, ulcerative colitis, psoriatic arthritis or seronegative spondyloarthropathy
* Other criteria to be reviewed by study doctor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLy (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (48):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calabasas, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brisbane, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
- Chile (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdivia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viña del Mar
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig, Germany
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kistarcsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucknow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
- Mexico (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chełm Śląski
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rimavska
- Ukraine (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivano-Frankivsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiev
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simferopol

REFERENCES:
- [Derived] Genovese MC, Lee E, Satterwhite J, Veenhuizen M, Disch D, Berclaz PY, Myers S, Sides G, Benichou O. A phase 2 dose-ranging study of subcutaneous tabalumab for the treatment of patients with active rheumatoid arthritis and an inadequate response to methotrexate. Ann Rheum Dis. 2013 Sep 1;72(9):1453-60. doi: 10.1136/annrheumdis-2012-202864. Epub 2013 Apr 18. PMID 23599435

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received a total of 6 subcutaneous (SC) injections (Weeks 0, 4, 8, 12, 16, and 20) of either placebo or 1 of 6 LY2127399 doses (1, 3, 10, 30, 60, or 120 milligrams [mg]) during the Treatment Phase. The Follow-up Phase took place Weeks 24-44 and the B-cell Follow-up Phase took place Weeks 44-72.
Groups:
- 1 mg LY2127399; 3 mg LY2127399; 10 mg LY2127399; 30 mg LY2127399; 60 mg LY2127399; 120 mg LY2127399: Administered SC every 4 weeks over a 24-week period (Weeks 0, 4, 8, 12, 16, and 20).
Period: Treatment Phase
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Started | 36 | 30 | 20 | 15 | 18 | 13 | 26
Completed | 33 | 25 | 17 | 15 | 16 | 13 | 23
Not Completed | 3 | 5 | 3 | 0 | 2 | 0 | 3
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 0 | 0 | 2
Not completed — Inadequate Response | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 1 | 0 | 0
Period: Follow-up Phases (Weeks 24-72)
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Started | 8 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.) | 8 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.) | 6 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.) | 4 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.) | 6 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.) | 0 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.) | 14 (Participants enrolling in an open-label extension study were not required to be in Follow-up Phase.)
Completed | 7 | 5 | 4 | 4 | 4 | 0 | 9
Not Completed | 1 | 3 | 2 | 0 | 2 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399 | Total
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 26 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (11.74) | 54.6 (11.67) | 53.4 (10.78) | 51.2 (13.78) | 54.5 (11.75) | 44.4 (13.83) | 50.7 (12.02) | 51.7 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 14 | 12 | 15 | 12 | 18 | 127
  Male | 6 | 4 | 6 | 3 | 3 | 1 | 8 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 25 | 22 | 13 | 8 | 11 | 5 | 17 | 101
  African | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Hispanic | 8 | 5 | 6 | 6 | 6 | 5 | 8 | 44
  East Asian | 2 | 2 | 1 | 0 | 1 | 3 | 1 | 10
  West Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 5
  Australia | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
  Chile | 4 | 2 | 2 | 2 | 3 | 2 | 2 | 17
  Germany | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hungary | 4 | 2 | 3 | 2 | 2 | 0 | 1 | 14
  India | 2 | 2 | 1 | 0 | 1 | 3 | 1 | 10
  Mexico | 5 | 4 | 4 | 2 | 3 | 3 | 4 | 25
  Poland | 12 | 8 | 5 | 4 | 4 | 2 | 5 | 40
  Romania | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 6
  Slovakia | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Ukraine | 5 | 3 | 3 | 2 | 2 | 0 | 8 | 23
  United States | 1 | 6 | 0 | 1 | 0 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 50 Response up to 24 Weeks
Description: ACR50 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis. An ACR50 Responder is defined as a participant with >50% improvement from baseline in both tender and swollen joint counts and in at least 3 of the following 5 criteria: physician global assessment, participant global assessment, functional ability measure (Health Assessment Questionnaire-Disability Index which measures participants' perceived degree of difficulty when performing various daily activities), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein.
Time Frame: Up to week 24
Population: Intent-to-treat (ITT) population included all randomized participants who received any amount of blinded study drug and who had at least 1 post-baseline efficacy assessment, Last Observation Carried Forward (LOCF). Two participants were excluded due to Good Clinical Practice (GCP) issues.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
percentage of participants | 18.1 | 17.7 | 17.0 | 15.0 | 11.8 | 11.8 | 37.0
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399 vs 3 mg LY2127399 vs 10 mg LY2127399 vs 30 mg LY2127399 vs 60 mg LY2127399 vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.059, Linear-quadratic regression model — This is p-value for the fitted ACR50 response rate and is based on the dose-response regression model and comes from the joint test of linear and quadratic dose response (response=dose+dose^2) from the likelihood ratio test
Statistical Analysis 2: Comparison: Placebo vs 1 mg LY2127399 vs 3 mg LY2127399 vs 10 mg LY2127399 vs 30 mg LY2127399 vs 60 mg LY2127399 vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.042, Linear-quadratic regression model — This is the p-value for the estimated dose level of the smallest dose, in milligrams (mg), that achieves at least 95% of the maximal efficacy (ED95) and is based on the comparisons that the ED95 yields a higher fitted response rate than placebo; This is ED95 in mg; ED95 = 119.0

2. Secondary Outcome: Percentage of Participants Achieving The American College of Rheumatology (ACR)20 Response up to 24 Weeks
Description: ACR20 Responder Index is composite of clinical, laboratory, and functional measures in rheumatoid arthritis. An ACR20 Responder is defined as participant with at least 20% improvement from baseline in both tender and swollen joint counts and in at least 3 of the following 5 criteria: physician global assessment, participant global assessment, functional ability measure (Health Assessment Questionnaire-Disability Index which measures participants' perceived degree of difficulty when performing various daily activities), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein.
Time Frame: Up to 24 weeks
Population: Intent-to-treat (ITT) population included all randomized participants who received any amount of blinded study drug and who had at least 1 post-baseline efficacy assessment, Last Observation Carried Forward (LOCF)/non-responder imputation (NRI). 2 participants were excluded due to Good Clinical Practice (GCP) issues.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo was administered subcutaneously (SC) every 4 weeks over a 24-week period.
- 1 mg LY2127399: 1 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
- 3 mg LY2127399: 3 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
- 10 mg LY2127399: 10 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
- 30 mg LY2127399: 30 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
- 60 mg LY2127399: 60 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
- 120 mg LY2127399: 120 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
percentage of participants | 43.2 | 43.6 | 44.3 | 46.9 | 53.5 | 61.5 | 70.1
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399 vs 3 mg LY2127399 vs 10 mg LY2127399 vs 30 mg LY2127399 vs 60 mg LY2127399 vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.044, Linear-quadratic regression model — This is the p-value for the fitted ACR20 response rate and is based on the dose-response regression model and comes from the joint test of linear and quadratic dose response (response=dose+dose^2) from the likelihood ratio test
Statistical Analysis 2: Comparison: Placebo vs 1 mg LY2127399 vs 3 mg LY2127399 vs 10 mg LY2127399 vs 30 mg LY2127399 vs 60 mg LY2127399 vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.005, Linear-quadratic regression model — This p-value is for estimated dose level of the smallest dose, in milligrams (mg), that achieves at least 95% of the maximal efficacy (ED95) of the ACR20 and is based on the comparisons that the ED95 yields a higher fitted response rate than placebo; This is the ED95 in mg; ED95 = 118.5

3. Secondary Outcome: Change From Baseline in the Tender Joint Count up to 24 Weeks
Description: Number of tender and painful joints was determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. Joints were assessed by pressure and joint manipulation on physical examination. Participant was asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both is translated into a single tender-versus-nontender dichotomy.
Time Frame: Baseline, up to 24 weeks
Population: Intent-to-treat (ITT) population included all randomized participants who received any amount of blinded study drug and who had at least 1 post-baseline efficacy assessment, Last Observation Carried Forward (LOCF). 2 participants were excluded due to Good Clinical Practice (GCP) issues.
Measure: Mean (Standard Deviation); unit: tender joints
Groups:
- 1 mg LY2127399: 1 milligram (mg) of LY2127399 was administered SC every 4 weeks over a 24-week period.
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
tender joints | -7.1 (8.21) | -7.3 (10.24) | -4.5 (7.74) | -8.7 (5.94) | -7.8 (7.68) | -7.4 (10.22) | -8.2 (6.41)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.623, ANCOVA — Pairwise comparison (2-sided) of 1 mg LY2127399 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.160, ANCOVA — Pairwise comparison (2-sided) of 3 mg LY2127399 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.568, ANCOVA — Pairwise comparison (2-sided) of 10 mg LY2127399 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.633, ANCOVA — Pairwise comparison (2-sided) of 30 mg LY2127399 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.754, ANCOVA — Pairwise comparison (2-sided) of 60 mg LY2127399 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.289, ANCOVA — Pairwise comparison (2-sided) of 120 mg LY2127399 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate

4. Secondary Outcome: Change From Baseline in Swollen Joint Count up to 24 Weeks
Description: The number of swollen joints was determined by examination of 28 joints which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
swollen joints | -5.6 (5.66) | -6.9 (6.10) | -5.7 (5.57) | -8.9 (6.03) | -5.4 (4.34) | -6.2 (6.19) | -7.3 (5.14)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.671, ANCOVA — Pairwise comparison (2-sided) of 1 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.696, ANCOVA — Pairwise comparison (2-sided) of 3 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.367, ANCOVA — Pairwise comparison (2-sided) of 10 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.645, ANCOVA — Pairwise comparison (2-sided) of 30 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.944, ANCOVA — Pairwise comparison (2-sided) of 60 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.133, ANCOVA — Pairwise comparison (2-sided) of 120 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate

5. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS) up to 24 Weeks
Description: DAS (modified to include the 28 joint count [DAS28]) consists of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP), and participant global assessment of his or her disease activity (participant global visual analog scale [pt global VAS]). The DAS28 is calculated by using the following formula: DAS28-CRP = 0.56*sqrt(28TJC) + 0.28*sqrt(28SJC) + 0.36*ln(CRP+1) + 0.014*pt global VAS + 0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 35 | 28 | 19 | 14 | 17 | 12 | 23
units on a scale | -1.448 (1.310) | -1.539 (1.346) | -1.026 (1.118) | -1.678 (0.987) | -1.536 (1.257) | -1.642 (1.222) | -1.915 (1.183)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.457, ANCOVA — Pairwise comparison (1-sided) of 1 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.874, ANCOVA — Pairwise comparison (1-sided) of 3 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.278, ANCOVA — Pairwise comparison (1-sided) of 10 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.357, ANCOVA — Pairwise comparison (1-sided) of 30 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.271, ANCOVA — Pairwise comparison (1-sided) of 60 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.048, ANCOVA — Pairwise comparison (1-sided) of 120 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as a covariate

6. Secondary Outcome: Percentage of Participants With A European League Against Rheumatism Responder Index Based on the 28 Joint Count (EULAR28) up to 24 Weeks
Description: The EULAR28 categorizes clinical response based upon improvement since baseline in the Disease Activity Score (DAS) modified to include the 28 joint count (DAS28) and post-baseline DAS28 level. DAS28 consists of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP), and participant global assessment of their disease activity (participant global visual analog scale [VAS]). EULAR28 categories include: No Response (improvement in DAS28 of less than or equal to 0.6 units or post-baseline DAS28 score greater than 5.1 with improvement by less than or equal to 1.2 units), Moderate Response (post-baseline DAS28 score less than or equal to 5.1 with improvement by more than 0.6 units but no greater than 1.2 units or post-baseline DAS28 score greater than 3.2 with improvement by more than 1.2 units), and Good Response (post-baseline DAS28 score less than or equal to 3.2 with improvement by more than 1.2 units).
Time Frame: Up to 24 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
percentage of participants
  Good response | 11.4 | 10.7 | 10.5 | 7.1 | 23.5 | 25.0 | 26.1
  Moderate response | 45.7 | 53.6 | 42.1 | 50.0 | 52.9 | 33.3 | 56.5
  No response | 42.9 | 35.7 | 47.4 | 42.9 | 23.5 | 41.7 | 17.4
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.875, Fisher Exact — This p-value is from 2-sided comparison of 1 mg LY2127399 versus placebo using Fisher's exact test for the 3 levels of EULAR response (good, moderate, no)
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 1.000, Fisher Exact — This p-value is from 2-sided comparison of 3 mg LY2127399 versus placebo using Fisher's exact test for the 3 levels of EULAR response (good, moderate, no)
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 1.000, Fisher Exact — This p-value is from 2-sided comparison of 10 mg LY2127399 versus placebo using Fisher's exact test for the 3 levels of EULAR response (good, moderate, no)
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.304, Chi-squared — This p-value is from a 2-sided comparison of 30 mg LY2127399 versus placebo using a Chi-square test for the 3 levels of EULAR response (good, moderate, no)
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.489, Chi-squared — This p-value is from a 2-sided comparison of 60 mg LY2127399 versus placebo using a Chi-square test for the 3 levels of EULAR response (good, moderate, no)
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.091, Chi-squared — This p-value is from a 2-sided comparison of 120 mg LY2127399 versus placebo using a Chi-square test for the 3 levels of EULAR response (good, moderate, no)

7. Secondary Outcome: Change From Baseline in the Participant's Assessment of Joint Pain up to 24 Weeks
Description: Participant's assessment of joint pain using a visual analog scale (VAS), which ranged from 0 to 100 mm, where 0 indicated no pain and 100 indicated worst possible pain.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
millimeters (mm) | -19.5 (27.50) | -17.8 (23.40) | -12.8 (19.76) | -21.2 (25.42) | -13.1 (21.95) | -17.6 (14.20) | -30.3 (25.93)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.746, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.393, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.549, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.619, ANCOVA — [p-value comment as in outcome 4, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.893, ANCOVA — [p-value comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.066, ANCOVA — [p-value comment as in outcome 4, analysis 6]

8. Secondary Outcome: Change From Baseline in the Participant's Assessment of Disease Activity up to 24 Weeks
Description: Participant's assessment of disease activity using a visual analog scale (VAS), which ranged from 0 to 100 mm, where 0 indicated no arthritis activity and 100 indicated extremely active arthritis.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 35 | 28 | 19 | 15 | 17 | 13 | 24
millimeters (mm) | -23.7 (24.76) | -21.2 (24.63) | -16.1 (18.58) | -22.5 (28.56) | -19.3 (17.58) | -15.5 (19.65) | -33.9 (22.68)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.583, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.311, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.752, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.737, ANCOVA — [p-value comment as in outcome 4, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.522, ANCOVA — [p-value comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.073, ANCOVA — [p-value comment as in outcome 4, analysis 6]

9. Secondary Outcome: Change From Baseline in the Physician's Assessment of Disease Activity up to 24 Weeks
Description: Physician's assessment of disease activity using a visual analog scale (VAS) that ranged from 0 to 100 mm, where 0 indicated no arthritis activity and 100 indicated extremely active arthritis.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
millimeters (mm) | -22.8 (22.02) | -22.8 (20.26) | -26.3 (26.09) | -30.2 (22.15) | -28.3 (20.62) | -21.4 (15.96) | -36.1 (17.06)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.969, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.352, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.406, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.266, ANCOVA — [p-value comment as in outcome 4, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.708, ANCOVA — [p-value comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.012, ANCOVA — [p-value comment as in outcome 4, analysis 6]

10. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) up to 24 Weeks
Description: Participant's assessment of physical function. Disability section of questionnaire scores participant's self-perception on degree of difficulty (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do) when dressing and grooming, arising, eating, walking, hygiene, reach, grip, and performing other daily activities. Scores for each of the functional areas were averaged to calculate the functional disability index. The HAQ-DI total score, which is the average of the nonmissing functional scores, ranges from 0 (no disability) to 3 (severe disability).
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
units on a scale | -0.281 (0.481) | -0.288 (0.609) | -0.206 (0.406) | -0.258 (0.373) | -0.292 (0.554) | -0.587 (0.546) | -0.370 (0.426)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.880, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.575, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.992, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.646, ANCOVA — [p-value comment as in outcome 4, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.054, ANCOVA — [p-value comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.472, ANCOVA — [p-value comment as in outcome 4, analysis 6]

11. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein (CRP) up to 24 Weeks
Description: Percent change = [(postbaseline CRP - baseline CRP)/baseline CRP]*100.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
percent change | 9.13 (136.683) | 18.28 (92.909) | 93.75 (265.331) | 5.60 (73.212) | 24.17 (188.146) | -34.42 (46.632) | 7.50 (132.313)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.952, ANCOVA — Pairwise comparison (2-sided) of 1 mg LY2123799 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable, treatment as the fixed factor, and the standardized rank baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.085, ANCOVA — Pairwise comparison (2-sided) of 3 mg LY2123799 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable, treatment as the fixed factor, and the standardized rank baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.143, ANCOVA — Pairwise comparison (2-sided) of 10 mg LY2123799 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable, treatment as the fixed factor, and the standardized rank baseline value as a covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.242, ANCOVA — Pairwise comparison (2-sided) of 30 mg LY2123799 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable, treatment as the fixed factor, and the standardized rank baseline value as a covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.317, ANCOVA — Pairwise comparison (2-sided) of 60 mg LY2123799 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable, treatment as the fixed factor, and the standardized rank baseline value as a covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.456, ANCOVA — Pairwise comparison (2-sided) of 120 mg LY2123799 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable, treatment as the fixed factor, and the standardized rank baseline value as a covariate

12. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness (FACIT) Fatigue Scale up to 24 Weeks
Description: The FACIT Fatigue Scale is a brief participant-reported measure of fatigue and consists of 13 items. Scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
units on a scale | 4.4 (12.22) | 3.9 (10.95) | 3.8 (8.04) | 8.1 (8.77) | 6.9 (8.08) | 8.0 (8.19) | 9.6 (7.83)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.833, ANCOVA — Pairwise comparison (2-sided) of 1 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as the covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.826, ANCOVA — Pairwise comparison (2-sided) of 3 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as the covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.091, ANCOVA — Pairwise comparison (2-sided) of 10 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as the covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.127, ANCOVA — Pairwise comparison (2-sided) of 30 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as the covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.243, ANCOVA — Pairwise comparison (2-sided) of 60 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as the covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.037, ANCOVA — Pairwise comparison (2-sided) of 120 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and the baseline value as the covariate

13. Secondary Outcome: Change From Baseline in the Short Form Health Survey (SF-36) up to 24 Weeks
Description: A self-reported questionnaire that consists of 36 questions covering 8 health domains (physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional, and general health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. The mental component summary (MCS) and the physical component summary (PCS) have been constructed based on the 8 SF-36 domains. MCS and PCS scores = 0 to 100 (higher scores indicate better health status).
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 17 | 13 | 24
units on a scale
  Physical Health Component | 4.284 (7.889) | 3.422 (7.592) | 2.534 (4.779) | 5.584 (7.905) | 3.680 (5.289) | 9.487 (8.366) | 4.053 (6.353)
  Mental Health Component | 3.623 (10.414) | 2.899 (13.094) | 4.263 (11.304) | 5.223 (11.289) | 4.166 (7.733) | 6.266 (7.139) | 9.198 (9.822)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.562, ANCOVA — P-value for physical health component. Pairwise comparison (2-sided) of 1 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.539, ANCOVA — P-value for physical health component. Pairwise comparison (2-sided) of 3 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.304, ANCOVA — P-value for physical health component. Pairwise comparison (2-sided) of 10 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.832, ANCOVA — P-value for physical health component. Pairwise comparison (2-sided) of 30 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value for physical health component. Pairwise comparison (2-sided) of 60 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.980, ANCOVA — P-value for physical health component. Pairwise comparison (2-sided) of 120 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 7: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.569, ANCOVA — P-value for mental health component. Pairwise comparison (2-sided) of 1 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 8: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.953, ANCOVA — P-value for mental health component. Pairwise comparison (2-sided) of 3 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 9: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.647, ANCOVA — P-value for mental health component. Pairwise comparison (2-sided) of 10 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 10: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.507, ANCOVA — P-value for mental health component. Pairwise comparison (2-sided) of 30 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 11: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.821, ANCOVA — P-value for mental health component. Pairwise comparison (2-sided) of 60 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate
Statistical Analysis 12: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.045, ANCOVA — P-value for mental health component. Pairwise comparison (2-sided) of 120 mg LY2123799 versus placebo using contrast statements within an analysis of covariance (ANCOVA) model with treatment as the fixed factor and baseline value as the covariate

14. Secondary Outcome: Pharmacokinetics of LY2127399: C-Trough Steady State Concentration at 24 Weeks
Description: C-trough is defined as the concentration of LY2127399 at the end of the dosing interval after the subcutaneous (sc) injection dosing once every 4 weeks. Mean C-trough value was obtained by conducting a simulation consisting of 1000 participants. The model was then used to predict the concentration-time profile at steady state. The pharmacokinetic (PK) parameters were then estimated from these concentration-time profiles.
Time Frame: 24 weeks
Population: The PK analysis population included all intent-to-treat (ITT) participants who received LY2127399 and who had evaluable PK data except 2 participants who were excluded due to Good Clinical Practice (GCP) issues.
Measure: Number; unit: micrograms per milliliter (µg/mL)
Groups:
- 120 mg of LY2127399: 120 mg of LY2127399 was administered SC every 4 weeks over a 24-week period.
Arm/Group | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg of LY2127399
Number analyzed (Participants) | 30 | 20 | 15 | 18 | 13 | 24
micrograms per milliliter (µg/mL) | 0.0100 | 0.0400 | 0.270 | 1.94 | 5.16 | 11.9

15. Secondary Outcome: Pharmacokinetics of LY2127399: T-Half Life (t1/2, Tau) at 24 Weeks
Description: T1/2,tau is defined as the apparent steady state elimination within the dosing interval. T1/2,tau was obtained by conducting a simulation consisting of 1000 participants. The model was then used to predict the concentration-time profile at steady state. The pharmacokinetic (PK) parameters were then estimated from these concentration-time profiles.
Time Frame: 24 weeks
Population: as for outcome 14
Measure: Number; unit: days
Arm/Group | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 30 | 20 | 15 | 18 | 13 | 24
days | 7.07 | 7.94 | 9.76 | 15.9 | 19.5 | 21.6

16. Secondary Outcome: Change From Baseline in the Absolute Total B Cell (CD20+CD3- Cells) Count up to 24 Weeks
Description: B-lymphocyte antigen CD20 or CD20 is an activated-glycosylated phosphoprotein expressed on the surface of all mature B-cells. Total B cell counts (CD20+CD3-) are represented by the number of cells per microliter (cells/µL). The reference range is 43 - 602 cells/µL.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 35 | 30 | 20 | 15 | 17 | 13 | 24
cells per microliter (cells/µL) | 17.63 (75.880) | -18.77 (96.410) | -50.85 (130.405) | -36.87 (71.287) | -68.59 (115.971) | -11.15 (111.577) | -27.88 (97.729)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.236, ANCOVA — Pairwise (2-sided) comparisons of 1 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable treatment as the fixed factor and the standardized rank baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.038, ANCOVA — Pairwise (2-sided) comparisons of 3 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable treatment as the fixed factor and the standardized rank baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.025, ANCOVA — Pairwise (2-sided) comparisons of 10 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable treatment as the fixed factor and the standardized rank baseline value as a covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.005, ANCOVA — Pairwise (2-sided) comparisons of 30 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable treatment as the fixed factor and the standardized rank baseline value as a covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.734, ANCOVA — Pairwise (2-sided) comparisons of 60 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable treatment as the fixed factor and the standardized rank baseline value as a covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.035, ANCOVA — Pairwise (2-sided) comparisons of 120 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with the standardized rank outcome variable treatment as the fixed factor and the standardized rank baseline value as a covariate

17. Secondary Outcome: Change From Baseline in Serum Immunoglobulin up to 24 Weeks
Description: Serum immunoglobulin measured by Immunoglobulin G (IgG), Immunoglobulin M (IgM), and Immunoglobulin A (IgA) levels.
Time Frame: Baseline, up to 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 24
gram per liter (g/L)
  IgG | -0.12 (2.964) | -0.14 (1.986) | -0.45 (3.179) | -0.45 (2.303) | -1.06 (2.650) | -0.93 (1.381) | -0.37 (2.147)
  IgM | 0.02 (0.323) | 0.07 (0.336) | -0.02 (0.269) | -0.11 (0.283) | -0.08 (0.531) | -0.30 (0.299) | -0.09 (0.384)
  IgA | -0.12 (0.482) | -0.09 (0.583) | -0.24 (0.712) | -0.53 (0.679) | -0.58 (0.977) | -0.42 (0.453) | -0.25 (0.631)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.901, ANCOVA — P-value for IgG. Pairwise comparison (2-sided) of 1 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.840, ANCOVA — P-value for IgG. Pairwise comparison (2-sided) of 3 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.882, ANCOVA — P-value for IgG. Pairwise comparison (2-sided) of 10 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.225, ANCOVA — P-value for IgG. Pairwise comparison (2-sided) of 30 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 5: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.340, ANCOVA — P-value for IgG. Pairwise comparison (2-sided) of 60 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 6: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.850, ANCOVA — P-value for IgG. Pairwise comparison (2-sided) of 120 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 7: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.447, ANCOVA — P-value for IgM. Pairwise comparison (2-sided) of 1 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 8: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.909, ANCOVA — P-value for IgM. Pairwise comparison (2-sided) of 3 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 9: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.152, ANCOVA — P-value for IgM. Pairwise comparison (2-sided) of 10 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 10: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.023, ANCOVA — P-value for IgM. Pairwise comparison (2-sided) of 30 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 11: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value for IgM. Pairwise comparison (2-sided) of 60 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 12: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value for IgM. Pairwise comparison (2-sided) of 120 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 13: Comparison: Placebo vs 1 mg LY2127399; Test type: Superiority or Other; p = 0.944, ANCOVA — P-value for IgA. Pairwise comparison (2-sided) of 1 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 14: Comparison: Placebo vs 3 mg LY2127399; Test type: Superiority or Other; p = 0.677, ANCOVA — P-value for IgA. Pairwise comparison (2-sided) of 3 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 15: Comparison: Placebo vs 10 mg LY2127399; Test type: Superiority or Other; p = 0.053, ANCOVA — P-value for IgA. Pairwise comparison (2-sided) of 10 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 16: Comparison: Placebo vs 30 mg LY2127399; Test type: Superiority or Other; p = 0.061, ANCOVA — P-value for IgA. Pairwise comparison (2-sided) of 30 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 17: Comparison: Placebo vs 60 mg LY2127399; Test type: Superiority or Other; p = 0.025, ANCOVA — P-value for IgA. Pairwise comparison (2-sided) of 60 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as the fixed factor, and standardized rank baseline value as a covariate
Statistical Analysis 18: Comparison: Placebo vs 120 mg LY2127399; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value for IgA. Pairwise comparison (2-sided) of 120 mg LY2127399 versus placebo using ranked analysis of covariance (ANCOVA) with standardized rank outcome variable, treatment as fixed factor, and standardized rank baseline value as a covariate

18. Secondary Outcome: Number of Participants Experiencing An Adverse Event
Description: Serious adverse events and other nonserious adverse events are located in the Reported Adverse Event section.
Time Frame: Baseline up to 24 weeks
Population: All randomized participants who received any amount of blinded study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399
Number analyzed (Participants) | 36 | 30 | 20 | 15 | 18 | 13 | 26
Participants
  Serious Adverse Events | 5 | 4 | 0 | 0 | 3 | 2 | 1
  Other Nonserious Adverse Events | 21 | 19 | 12 | 9 | 11 | 8 | 13

ADVERSE EVENTS:
Groups:
- Placebo - Follow-up Period; 1 mg LY2127399 - Follow-up Period; 3 mg LY2127399 - Follow-up Period; 10 mg LY2127399 - Follow-up Period; 30 mg LY2127399 - Follow-up Period; 60 mg LY2127399 - Follow-up Period; 120 mg LY2127399 - Follow-up Period: Participants were assessed but did not receive any study medication during the follow-up period.
Arm/Group | Placebo | 1 mg LY2127399 | 3 mg LY2127399 | 10 mg LY2127399 | 30 mg LY2127399 | 60 mg LY2127399 | 120 mg LY2127399 | Placebo - Follow-up Period | 1 mg LY2127399 - Follow-up Period | 3 mg LY2127399 - Follow-up Period | 10 mg LY2127399 - Follow-up Period | 30 mg LY2127399 - Follow-up Period | 60 mg LY2127399 - Follow-up Period | 120 mg LY2127399 - Follow-up Period
Serious Adverse Events (participants affected / at risk) | 5/36 | 4/30 | 0/20 | 0/15 | 3/18 | 2/13 | 1/26 | 0/8 | 0/8 | 1/6 | 0/4 | 1/6 | 0/0 | 0/14
Other Adverse Events (participants affected / at risk) | 21/36 | 19/30 | 12/20 | 9/15 | 11/18 | 8/13 | 13/26 | 1/8 | 2/8 | 1/6 | 3/4 | 3/6 | 0/0 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | 1 mg LY2127399 (N=30) | 3 mg LY2127399 (N=20) | 10 mg LY2127399 (N=15) | 30 mg LY2127399 (N=18) | 60 mg LY2127399 (N=13) | 120 mg LY2127399 (N=26) | Placebo - Follow-up Period (N=8) | 1 mg LY2127399 - Follow-up Period (N=8) | 3 mg LY2127399 - Follow-up Period (N=6) | 10 mg LY2127399 - Follow-up Period (N=4) | 30 mg LY2127399 - Follow-up Period (N=6) | 60 mg LY2127399 - Follow-up Period (N=0) | 120 mg LY2127399 - Follow-up Period (N=14)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | 1 mg LY2127399 (N=30) | 3 mg LY2127399 (N=20) | 10 mg LY2127399 (N=15) | 30 mg LY2127399 (N=18) | 60 mg LY2127399 (N=13) | 120 mg LY2127399 (N=26) | Placebo - Follow-up Period (N=8) | 1 mg LY2127399 - Follow-up Period (N=8) | 3 mg LY2127399 - Follow-up Period (N=6) | 10 mg LY2127399 - Follow-up Period (N=4) | 30 mg LY2127399 - Follow-up Period (N=6) | 60 mg LY2127399 - Follow-up Period (N=0) | 120 mg LY2127399 - Follow-up Period (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
H1n1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichophytic granuloma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt interval abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical diathermy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days